CLINICAL TRIAL: NCT03270176
Title: A Phase-Ib Dose-Finding Study of the SMAC Mimetic Debio 1143 When Given in Combination With the Anti-PD-L1 Antibody Avelumab to Patients With Advanced Solid Malignancies and, in an Expansion Cohort, to Patients With Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) After Platinum-Based Therapy
Brief Title: A Dose-Finding Study of the Second Mitochondrial Activator of Caspases (SMAC) Mimetic Debio 1143 When Given in Combination With Avelumab to Participants With Advanced Solid Malignancies and to Participants With Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) After Platinum-Based Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Debio 1143-NSCLC-105; 2018-000494-71 (EudraCT Number)
Record Dates: First submitted 2017-08-29; First posted 2017-09-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — N-benzhydryl-5-(2-(methylamino)propanamido)-3-(3-methylbutanoyl)-6-oxodecahydropyrrolo(1,2-a)(1,5)diazocine-8-carboxamide; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Debio 1143 and Avelumab (Experimental): Part A: Participants will receive Debio 1143 100 to 250 milligram (mg) capsule orally at an escalating dose levels for 10 days every 2 weeks along with avelumab 10 milligrams per kilogram (mg/kg) as an intravenous (IV) infusion every 2 weeks.
  Part B: Participants will receive Debio 1143 capsules orally at a recommended phase 2 dose (RP2D) of 200 mg/day (days 1-10 and 15-24 every 28 days ([q4w]) in combination with avelumab IV infusion at the standard dose unless disease progression or unacceptable toxicity occurs, as judged by investigators up to 26 cycles (each cycle is of 28 days).
  Interventions: Drug: Debio 1143; Drug: Avelumab

INTERVENTIONS:
Drug: Debio 1143 — Debio 1143 100 to 250 mg, capsule orally for 10 days every 2 weeks.
Drug: Avelumab — Avelumab 10 mg/kg intravenous infusion every 2 weeks.

SUMMARY:
The study is primarily designed to assess the safety and tolerability of escalating oral doses of Debio 1143 and preliminary anti-tumour activity when combined with the standard dose of avelumab in participants with advanced solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

Part A • With advanced solid malignancies who are not eligible for standard therapy or for whom standard therapy has failed

Part B

• With histologically or cytologically confirmed NSCLC of stage IIIB or IV (per 7th International Association for the Study of Lung Cancer classification) that has progressed after one line of platinum containing doublet chemotherapy

Part A and B

* Willingness and feasibility to provide a tumor biopsy sample both at screening and during treatment (If archived tumor material not older than 1 year is available, then the screening biopsy will not be performed).
* Participants with prior radiation therapy must have measurable disease in non-irradiated sites or documented evidence of progression within the radiation field.
* With known central nervous system (CNS) must have completed primary brain therapy (such as whole brain radiotherapy, stereotactic radiosurgery, or complete surgical resection) and must have remained clinically stable, asymptomatic, and without steroid treatment for at least 21 days.

Exclusion Criteria:

* Not recovered (i.e. toxicity grade >1) from prior investigational drug and/or anti-cancer therapy (chemo- or palliative radiotherapy).
* Symptomatic and/or progressive brain metastasis or carcinomatous meningitis.
* Immunosuppressive agents (such as steroids) for any reason should be tapered off before initiation of study treatment (except low-dose prednisone at a total dose of up to 10 mg/day).

Part B only

* Tumor activating epidermal growth factor receptor (EGFR) mutation(s) or anaplastic lymphoma kinase (ALK)/ROS1 translocation/rearrangement (testing required in non-squamous participants if status is unknown).
* More than one prior line of chemotherapy and one line of anti-PD1/PDL1 therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Part A: Maximum Tolerated Dose (MTD) | Baseline up to Cycle 1 (4 Weeks)
  MTD:dose with estimated probability of dose limited toxicity(DLT) below 30%.DLT:any of following adverse events(AEs) during 1st treatment cycle if deemed related to treatment:grade (gr) 3/4 febrile neutropenia/any gr 4 neutropenia of >5 days duration;gr 4 thrombocytopenia[<25000 per cubic millimetre(/mm^3)]/gr 3(<50000/mm^3),associated with medically concerning bleeding;gr ≥3 non-hematologic laboratory value;non-hematologic toxicity of gr 3/4,gr ≥2 uveitis/eye pain that does neither respond to topical therapy nor abate to gr 1within the avelumab re-treatment period/that required systemic treatment;gr ≥2 pneumonitis/interstitial lung disease that not resolve with dose delay and systemic steroids;toxicity related to study drug that requires dosing delay of >2weeks,dose reduction,premature discontinuation of any of two;other drug related AE in the opinion of investigator is of potential clinical significance so that further dose-escalation would expose participants to unacceptable risk.
Part B: Objective Response Rate (ORR) | From first occurrence of objective response until disease progression or death from any cause or switch to a new systemic therapy or end of study (Up to 2 years)
  Objective response is defined as any partial response (PR) or complete response (CR) recorded from the start of study treatment until disease progression/recurrence is documented, a new systemic therapy is started or analysis cut-off, whichever occurs first. It is assessed by using Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1. RECIST v1.1 criteria- CR: disappearance of all target lesions, any pathological lymph nodes must have reduction in short axis to <10 millimeter (mm). PR: At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameter.

SECONDARY OUTCOMES:
Part A and B: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to 90 days after the last dose of study drug (up to 2.5 years)
  An AE is any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. An SAE is any untoward medical occurrence at any dose that results in death; is life-threatening; requires hospitalization; results in persistent or significant disability or in congenital anomaly/birth defect. Severity will be graded by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.03.
Part A and B: Change in Tumor Size | Day 1 of cycle 3 up to 6 months; Day 1 of cycle 9, 12, 15, 18, 21, 24, 26 or until disease progression/EOT (up to 2 years)
  Change in tumor size is the maximum reduction or, in case of no reduction, the minimum increase in tumor size from the start of study treatment until disease progression/recurrence, the start of a new systemic therapy or analysis cut-off, whichever occurs first.
Part A and B: Objective Response Rate | At the end of Cycle 6 (168 days)
  Objective response is defined as any PR or CR recorded from the start of study treatment until disease progression/recurrence is documented, a new systemic therapy is started or analysis cut-off, whichever occurs first. It is assessed by using RECIST criteria. CR: disappearance of all target lesions, any pathological lymph nodes must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameter.
Part A and B: Best Overall Response (BOR) | Day 1 of cycle 3 up to 6 months; Day 1 of cycle 9, 12, 15, 18, 21, 24, 26 or until disease progression/EOT (up to 2 years)
  Best overall response (BOR) is defined as the best response (CR, PR, stable disease or disease progression) recorded from the start of study treatment until disease progression/recurrence is documented, a new systemic therapy is started or analysis cut-off, whichever occurs first. It is assessed by using RECIST criteria version 1.1. CR: disappearance of all target lesions, any pathological lymph nodes must have reduction in short axis to <10 millimeter (mm). PR: At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameter. Disease progression: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). Stable Disease: Neither sufficient shrinkage to qualify for PR, nor sufficient increase to qualify for disease progression, taking as reference the smallest sum diameter while on study.
Part A and B: Duration of Response | Baseline up to Cycle 26 (2 years) or until disease progression/EOT
  Duration of response is the time from documentation of tumor response to disease progression was observed in participants with CR or PR. RECIST v1.1 criteria- CR: disappearance of all target lesions, any pathological lymph nodes must have reduction in short axis to <10 millimeter (mm). PR: At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameter. Disease progression: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Part A and B: Disease Control Rate | Day 1 of cycle 3 up to 6 months; Day 1 of cycle 9, 12, 15, 18, 21, 24, 26 or until disease progression/EOT (up to 2 years)
  Disease control is derived as CR, PR or stable disease lasting at least 16 weeks reported during the study. RECIST v1.1 criteria- CR: Disappearance of all target lesions, any pathological lymph nodes must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameter.
Part A and B: Progression Free Survival (PFS) | Up to 6 months, 1 and 2 years of treatment initiation
  PFS duration is defined as the time elapsed between treatment initiation and tumor progression or death from any cause, whichever occurs first. RECIST v1.1 criteria- CR: disappearance of all target lesions, any pathological lymph nodes must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameter. Disease progression: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Part A and B: Overall Survival (OS) | Up to 6 months, 1 and 2 years of treatment initiation
  OS is defined as the time elapsed between treatment initiation and death from any cause.
Part A and B: Assessment of Pharmacokinetic Parameters | Up to Cycle 25 (700 days)

CONTACTS AND LOCATIONS:
Locations (9):
- Canada (4):
  - Cross Cancer Center Dept Medicine, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - The Ottawa Hospital Cancer Centre (TOHCC), Ottawa, Ontario
- Poland (3):
  - Instytut Medyczny Santa Familia Sp. z o. o., Lodz
  - Med-Polonia Sp. z o.o., Ulica Obornicka, Poznan
  - Wojewódzki Szpital Zespolony im. Ludwika Rydygiera, Torun
- Romania (2):
  - Institutul Oncologic "Prof. Dr. Ion Chiricuţă" Cluj Napoca, Cluj-Napoca
  - Centrul de Oncologie, S.C. Centrul de Oncologie Sf. Nectarie S.R.L, Oncologie Medicala, Craiova

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goss G, Ciuleanu T, Ramlau R, Renouf DJ, Chu Q, Kalinka E, Sawrycki P, Bramson J, Nelson BH, Crabbe R, LaCasse E, Lo B, Sahlender DA, Crompton P, Brichory F, Piggott L, Schenker M, Juergens R. Xevinapant plus avelumab in advanced solid tumours, with a dose expansion in advanced non-small-cell lung cancer: exploratory biomarker, safety and efficacy analyses from an open-label, nonrandomised phase Ib study. Ther Adv Med Oncol. 2025 May 8;17:17588359251332154. doi: 10.1177/17588359251332154. eCollection 2025. PMID 40351326